CLINICAL TRIAL: NCT00630149
Title: Open-Label Single-Arm Phase 2 Study of Alimta in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma Who Have Had Prior Platinum Based Chemotherapy
Brief Title: Study of Alimta in Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC) Who Have Had Prior Platinum Based Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H3E-GH-0034
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Nasopharyngeal Neoplasms; Pemetrexed
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — Pemetrexed

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Pemetrexed (Alimta)

INTERVENTIONS:
Drug: Pemetrexed (Alimta) — 500 mg/m2 in Cycle 1, every 3 weeks, with folic acid and vitamin B12 supplementation.
  Other Names: Alimta

SUMMARY:
This is a pilot phase II study of locally advanced or metastatic nasopharyngeal carcinoma (NPC) with the single drug Alimta. The objective of this study is to assess efficacy and safety profiles of Alimta as 2nd line treatment for patients with advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of nasopharyngeal carcinoma.
* Locally recurrent or metastatic disease.
* Patients must have previously received one platinum based chemotherapy regimen for palliative therapy of locally advanced or metastatic disease.
* Prior platinum based chemotherapy completed at least 3 months prior to study enrollment and the patient must have recovered from toxic effects of the treatment.
* Previous radiation therapy is allowed, but should have been limited and must not have included whole pelvis radiation. Patients must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed 30 days before study entry. Lesions that have been radiated cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.
* Disease status must be that of measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Scale.
* Estimated life expectancy of at least 8 weeks.
* Patient compliance and geographic proximity that allow adequate follow-up.
* Adequate organ function including the following: Bone marrow: absolute neutrophil count (ANC) >or= 1.5x10^9/L, platelets >or= 100x10^9/L, hemoglobin >or= 9g/dL. Hepatic: bilirubin <1.5 x ULN, alkaline phosphatase, aspartate transaminase (AST) and alanine transaminase (ALT) < 2.5 x ULN (alkaline phosphatase, AST, ALT < 5 x ULN is acceptable if liver has tumor involvement). Renal: calculated creatinine clearance > 45 ml/min.
* Men or women of at least 18 years of age.
* For women: Must be surgically sterile, post-menopausal, or compliant with a medically approved contraceptive regimen during and for 3 months after the treatment period; must have a negative serum or urine pregnancy test and must not be lactating. For men: Must be surgically sterile, or compliant with a contraceptive regimen during and for 3 months after the treatment period.
* Signed informed consent from patient.

Exclusion Criteria:

* Known or suspected brain metastasis. Patients who have clinical signs or symptoms that are suspicious of brain metastasis must have a pretreatment computed tomography (CT) or magnetic resonance imaging (MRI) of the brain. A patient with documented brain metastasis, at the time of consideration for study entry or in the past, will be excluded from entering in the study.
* Have previously completed or withdrawn from this study, or received Alimta previously outside this study.
* Concurrent administration of any other tumor therapy.
* Active infection (at the discretion of the investigator).
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Pregnancy or breast feeding.
* History of significant neurological or mental disorder, including seizures or dementia.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Inability to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs) 2 days before, the day of, and 2 days after the dose of Alimta. If a patient is taking a NSAID (Cox-2 inhibitors included) or salicylate with a long half-life, it should not be taken 5 days before, the day of, and 2 days after the dose of Alimta.
* Presence of clinically relevant third-space fluid collections that cannot be controlled by drainage or other procedures prior to study entry.
* Inability or unwillingness to take folic acid, vitamin B12 supplementation, or dexamethasone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
response rate | Jan 2010

SECONDARY OUTCOMES:
progression-free survival | Jan 2010
overall survival | Jan 2010
safety profile of pemetrexed (Alimta) treatment | Jan 2010
pharmacokinetic analysis of half-life, maximum plasma concentration (Cpmax), clearance (CL), area under the curve (AUC), and apparent volume of distribution | Jan 2010
evaluate the relationship between the expression of alpha folate receptor protein, TS and clinical response | Jan 2010

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — Cancer Center of Sun-Yat Sen University (CCSYSU)
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China